CLINICAL TRIAL: NCT01541553
Title: A Sequential Treatment Regimen of Cryotherapy and Picato® for the Treatment of Actinic Keratosis on the Face and Scalp
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0041-21
Record Dates: First submitted 2012-02-17; First posted 2012-03-01 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2016-07

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEP005 Gel, 0.015% (Active Comparator): Cryotherapy followed by PEP005 Gel, 0.015%
  Interventions: Procedure: Cryotherapy; Drug: Ingenol metabute
- Vehicle gel (Placebo Comparator): Cryotherapy followed by vehicle gel
  Interventions: Procedure: Cryotherapy; Drug: Vehicle

INTERVENTIONS:
Procedure: Cryotherapy — Cryotherapy of all visible AKs (4-8 lesions, "baseline lesions") in the selected treatment area
Drug: Vehicle — Field treatment with vehicle gel once daily for 3 consecutive days.
  Arms: Vehicle gel
Drug: Ingenol metabute — Field treatment with vehicle gel once daily for 3 consecutive days.
  Other Names: Picato® gel, 0.015%
  Arms: PEP005 Gel, 0.015%

SUMMARY:
The purpose of this trial is to compare the rate of complete clearance of actinic keratosis (AK) using sequential cryotherapy and field treatment with PEP005 Gel compared to cryotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be competent to understand the nature of the trial and provide informed consent.
* Subjects with 4 to 8 clinically typical, visible and discrete AKs within a contiguous 25 cm2 treatment area on the face or scalp.
* Subject at least 18 years of age.
* Female subjects must be of either:

  * Non-childbearing potential, i.e. post-menopausal or have a confirmed clinical history of sterility (e.g. the subject is without a uterus) or,
  * Childbearing potential, provided there is a confirmed negative urine pregnancy test prior to study treatment, to rule out pregnancy.
* Female subjects of childbearing potential must be willing to use effective contraception.

Exclusion Criteria:

* Location of the selected treatment area:

  * on any location other than the face or scalp
  * within 5 cm of an incompletely healed wound
  * within 10 cm of a suspected basal cell carcinoma (BCC) or SCC
* Prior treatment with PEP005 Gel on face or scalp.
* Selected treatment area lesions that have:

  * atypical clinical appearance and/or
  * recalcitrant disease
* History or evidence of skin conditions other than the trial indication that would interfere with evaluation of the trial medication
* Clinical diagnosis/history or evidence of any medical condition that would expose a subject to an undue risk of a significant AE or interfere with assessments of safety and efficacy.
* Any abnormal vital signs measurements that are medically significant or would impact the safety of the subject or the interpretation of the trial results.
* Anticipated need for hospitalization or out-patient surgery during the first 15 days after the first trial medication application.
* Known sensitivity or allergy to any of the ingredients in PEP005 Gel
* Recent excessive exposure to ultraviolet light
* Current enrolment or participation in a clinical trial within 30 days of entry into this study
* Subjects previously randomised in the trial
* Female subjects who are breastfeeding

Prohibited Therapies and/or Medications within 2 weeks prior to Visit 1

* Cosmetic or therapeutic procedures within 2 cm of the selected treatment area
* Use of acid-containing therapeutic products within 2 cm of the selected treatment area
* Use of topical medicated creams, ointments, lotions, gels, foams or sprays

Prohibited Therapies and/or Medications: within 4 weeks prior to visit 1:

* Treatment with immunomodulators, cytotoxic drugs or inter-feron /interferon inducers
* Treatment with systemic medications that suppress the immune system
* Treatment/therapy with ultraviolet light A (UVA) or ultraviolet light B (UVB).

Prohibited Therapies and/or Medications within 8 weeks prior to visit 1:

* Treatment with 5-FU, imiquimod, diclofenac sodium, or photodynamic therapy: within 2 cm of the selected treatment area.

Prohibited Therapies and/or Medications within 6 months prior to visit 1

* Use of systemic retinoids or biologic / mono-clonal antibody therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Berman, MD, Ph.D, Principal Investigator
Locations (35):
- United States (35):
  - Center for Dermatology Clinical Research, Fremont, California
  - Dermatology Specialists, Inc., Oceanside, California
  - Skin Surgery Medical Group, Inc., San Diego, California
  - University Clinical Trials, Inc., San Diego, California
  - Colorado Medical Research Center, Inc., Denver, Colorado
  - About Skin Dermatology and DermSurgery, PC, Englewood, Colorado
  - The Center for Clincial and Cosmetic Research, Aventura, Florida
  - Study Protocol, Inc., Boynton Beach, Florida
  - North Florida Dermatology Associates, PA, Jacksonville, Florida
  - University of South Florida, Carol and Frank Morsani Center for Advanced Healthcare, Tampa, Florida
  - MedaPhase, Newnan, Georgia
  - Gwinnett Clinical Research Center, Inc., Snellville, Georgia
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Laser & Skin Surgery Center of Indiana, Carmel, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Great Lakes Research Center, Bay City, Michigan
  - Henry Ford Medical Centre - New Center One, Department of Dermatology, Detroit, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Mount Sinai School of Medicine, New York, New York
  - Skin Search of Rochester, Inc., Rochester, New York
  - Long Island Skin Cancer and Dermatologic Surgery, Smithtown, New York
  - Oregon Medical Research Center, PC, Portland, Oregon
  - Oregon Health & Science University, Dept. of Dermatology, Portland, Oregon
  - Philadelphia Institute of Dermatology, Fort Washington, Pennsylvania
  - Dermatology Research Associates, Inc., Nashville, Tennessee
  - Arlington Research Center, Inc., Arlington, Texas
  - Suzanne Bruce and Associates, P.A., Houston, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - The Education & Research Foundation, Inc., Lynchburg, Virginia
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Premier Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berman B, Goldenberg G, Hanke CW, Tyring SK, Werschler WP, Knudsen KM, Larsson T, Swanson N. Efficacy and safety of ingenol mebutate 0.015% gel after cryosurgery of actinic keratosis: 12-month results. J Drugs Dermatol. 2014 Jun;13(6):741-7. PMID 24918567
- [Derived] Berman B, Goldenberg G, Hanke CW, Tyring SK, Werschler WP, Knudsen KM, Goncalves J, Larsson T, Skov T, Swanson N. Efficacy and safety of ingenol mebutate 0.015% gel 3 weeks after cryosurgery of actinic keratosis: 11-week results. J Drugs Dermatol. 2014 Feb;13(2):154-60. PMID 24509965
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 367 subjects were enrolled of whom 38 were screen failures. The remaining 329 subjects were randomised at Visit 1.
Groups:
- PEP005 Gel, 0.015%: Cryotherapy followed by PEP005 Gel, 0.015%
  Cryotherapy of all visible AKs (4-8 lesions, "baseline AKs") in the selected treatment area, 2-4 weeks healing time followed by field treatment with PEP005 gel, 0.015% once daily for 3 consecutive days
- Vehicle Gel: Cryotherapy followed by vehicle gel
  Cryotherapy of all visible AKs (4-8 lesions, "baseline AKs") in the selected treatment area, 2-4 weeks healing time followed by field treatment with vehicle gel once daily for 3 consecutive days.
Period: Overall Study
Arm/Group | PEP005 Gel, 0.015% | Vehicle Gel
Started | 167 | 162
Completed | 155 | 148
Not Completed | 12 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEP005 Gel, 0.015% | Vehicle Gel | Total
Number analyzed (Participants) | 167 | 162 | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (9.4) | 67.4 (9.3) | 67 (9.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 61 | 133
  >=65 years | 95 | 101 | 196
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 138 | 133 | 271
Region of Enrollment [Number; unit: participants]
  United States | 167 | 162 | 329

OUTCOME MEASURES:

1. Primary Outcome: Complete Clearance of AKs at Week 11
Description: To determine the 11-week rate of complete clearance of AKs (defined as no clinically visible AKs) in the selected treatment area using sequential cryotherapy and field treatment with PEP005 Gel compared to cryotherapy alone.
Time Frame: 11 weeks
Measure: Number; unit: participants
Arm/Group | PEP005 Gel, 0.015% | Vehicle Gel
Number analyzed (Participants) | 167 | 162
participants | 101 | 80

2. Secondary Outcome: Percentage Change From Baseline in Number of AKs at Week 11
Description: Percentage change from baseline in number of AKs at Week 11
Time Frame: Baseline to week 11
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | PEP005 Gel, 0.015% | Vehicle Gel
Number analyzed (Participants) | 167 | 162
percentage of change | 81.1 (31.8) | 74.1 (34.4)

3. Secondary Outcome: Partial Clearance of AKs at Week 11
Description: Partial clearance of AKs at Week 11, defined as 75% or greater reduction from baseline in the number of clinically visible AKs in the selected treatment area at Week 11
Time Frame: Week 11
Measure: Number; unit: participants
Arm/Group | PEP005 Gel, 0.015% | Vehicle Gel
Number analyzed (Participants) | 167 | 162
participants | 130 | 109

ADVERSE EVENTS:
Arm/Group | PEP005 Gel, 0.015% | Vehicle Gel
Serious Adverse Events (participants affected / at risk) | 7/167 | 4/162
Other Adverse Events (participants affected / at risk) | 0/167 | 0/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEP005 Gel, 0.015% (N=167) | Vehicle Gel (N=162)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischeamic (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor is entitled to review and comment on publications prior to submission or presentation.

Upon request of the sponsor, the investigator shall delay publication or presentation to allow for protection of the sponsors inventions and other intellectual property.